CLINICAL TRIAL: NCT04634032
Title: Gene Expression and DNA Variation Analysis of Sacs to Identify the Pathophysiology of Indirect Inguinal Hernia
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Oguz Kizilkaya, Resident, Trakya University
Other Study IDs: HerniaOK
Record Dates: First submitted 2020-11-02; First posted 2020-11-18 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Indirect Inguinal Hernia; Genetic Predisposition to Disease
Keywords: indirect inguinal hernia; GATA6; TBX3; SNP; gene expression
MeSH Terms: conditions — Hernia, Inguinal; Genetic Predisposition to Disease | interventions — Gene Expression; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 14 Days
Biospecimen Retention: Samples With DNA — Patent processus vaginalis and preputial tissue samples for mRNA expression analysis, peripheral white blood cells for SNP analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hernia: Patients planned to undergo routine indirect inguinal hernia repair procedure
  Interventions: Genetic: mRNA expression and SNP analysis; Diagnostic Test: Blood sampling
- Control: Patients planned to undergo routine circumcision procedure
  Interventions: Genetic: mRNA expression and SNP analysis; Diagnostic Test: Blood sampling

INTERVENTIONS:
Genetic: mRNA expression and SNP analysis — mRNA expression and SNP analysis from samples
Diagnostic Test: Blood sampling — Peripheral blood sampling for SNP analysis

SUMMARY:
The aim of the project is to show that gene expression levels change in at least one of the GATA6 and T-box transcription factor 3 (TBX3) genes in indirect inguinal hernia sacs, thus revealing that this pathway causes an error in the sac closure pathway.

Indirect inguinal hernia is an important condition for human health as it is common in the community and can lead to life-threatening or permanent loss of function. In addition, since the treatment is performed surgically, the follow-up and treatment process of the patients should be managed carefully in terms of complications and costs. By explaining the mechanisms of the occurrence of this disease, important steps will be taken in terms of both human health and the development of science. Moreover, the data to be collected may open new horizons in the treatment of inguinal hernia.

20 inguinal hernia patients those consecutively applied to Trakya University Medical Faculty Department of Pediatric Surgery and 20 circumcision patients as control group will be included in the study.

DETAILED DESCRIPTION:
Indirect inguinal hernia is one of the pathologies that is widely researched in national and international studies because of its high prevalence in the community and its life-threatening or permanent loss of function. However, no point has been reached regarding the etiology of this disease and a consensus has been reached.

The investigators believe that the study will contribute to the explanation of the formation mechanisms of the mentioned disease. Considering the high prevalence of this disease and its potential for life-threatening, the investigators anticipate that the analysis of the relevant genes for the Turkish population will make significant contributions to the public health. In the literature, analysis of GATA6 SNPs in the Chinese population has subsequently associated certain polymorphisms with indirect inguinal hernia. It is also been stated that TBX3 gene pathologies may be associated with inguinal hernia.

However, there is no study in the literature about the patent processus vaginalis expression levels of these genes. There is no study on the SNP analysis of these genes in Turkish population. For these reasons, the first time the expression / SNP analysis of the specified genes in Turkish society will be carried out will make an additional contribution to scientific knowledge. As stated clearly in the studies, the implementation of medical treatment of indirect inguinal hernia may change the approach of the pediatric surgical community to indirect inguinal hernia. In order for medical treatment to be carried out, the formation pathways and genetic origins of the disease must be clearly revealed.

Investigating the relationship of GATA6 and TBX3 genes, which are known to be involved in connective tissue homeostasis, with the mechanisms of indirect inguinal hernia formation, will contribute to the studies in the literature and is important in terms of revealing whether the treatment of these diseases can be performed medically in the future.

The study aims to reveal that gene expression levels in indirect inguinal hernia sacs due to SNPs in at least one of the GATA6 and TBX3 genes, thus causing an error in the sac closure pathway. The hypothesis of the study; It is stated that the gene expression levels of at least one of GATA6 and TBX3 in the sacs of inguinal hernia patients are altered.

The primary goal of this study is; To determine the level of GATA6 and TBX3 gene expression in sacs obtained from indirect inguinal hernia patients. The secondary goal is to investigate SNPs in the leukocytes of these patients and to investigate whether the genetic elements in our hypothesis in these diseases are regulated by different genes acting as transcription factors.

Considering that indirect inguinal hernia poses significant health risks, especially in children, it is predicted that the results to be obtained may contribute to clarification of the etiology and non-invasive methods other than surgery.

ELIGIBILITY:
Inclusion Criteria:

* to accept to participate the study
* pediatric age
* isolated indirect inguinal hernia patient with no additional systemic/congenital disease
* patients requesting circumcision procedure with no additional systemic/congenital disease

Exclusion Criteria:

* patients with any syndromic disease
* patients with hypospadias
* patients with undescended testes
* patients with umbilical hernia

Max Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Indirect inguinal hernia development differs between both sexes , our study aims to research indirect inguinal hernia in male population
Study Population: All patients applied to the Trakya University Hospital Pediatric Surgery Clinic that meet the inclusion criteria and whose legal representative gave consent to be enrolled included to the study.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2019-10-22 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2020-11-20 (Estimated)

PRIMARY OUTCOMES:
Gene expression and Single Nucleotide Polymorphism analysis | up to 3 months after completion of the study
  Determining the varieties of messenger ribonucleic acid (mRNA) expression levels between groups and possible Single Nucleotide Polymorphisms (SNP)

CONTACTS AND LOCATIONS:
Overall Officials: Oguz Kizilkaya, Principal Investigator — Trakya University
Locations (1):
- Trakya University, Edirne, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is no plan to share the data at this time but it may be possible after completion of the publication process.